CLINICAL TRIAL: NCT06250777
Title: A Phase 2 Trial to Assess Efficacy and Safety of T-DXd in HER2-mutant Advanced Lung Cancer Patients With Asymptomatic Brain Metastases.
Brief Title: Efficacy and Safety of T-DXd in HER2-mutant Advanced Lung Cancer Patients With Asymptomatic Brain Metastases
Acronym: ELPIS
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Chang Gon Kim, Principal Investigator, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1364
Record Dates: First submitted 2024-01-21; First posted 2024-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer(NSCLC); Human epidermal growth factor receptor 2 (HER-2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab Deruxtecan (Experimental)
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Chemotherapy : Every 3weeks as below until withdrawal of patient consent, progression, death or loss to follow-up:
  - Trastuzumab Deruxtecan (T-DXd) 5.4mg/kg

SUMMARY:
'1. Objective

* Primary objective

  - Median Intracranial Progression-free survival(icPFS) as defined by RANO(Response Assessment in Neuro-Oncology) criteria
* Secondary objective

  * Progression free survival(PFS) as defined by RECIST 1.1
  * Median Intracranial progression free survival(icPFS) as defined by RECIST 1.1
  * Intracranial objective response rate(icORR) as defined by RECIST 1.1
  * Overall response rate(ORR) as defined by RECIST 1.1
  * Duration of response(DoR) as defined by RECIST 1.1
  * Disease control rate (DCR) defined by RECIST 1.1
  * Overall survival (OS) ; The time from the date of inital IP administration to death due to any cause
  * Pattern of Progression ; Site of next progression
* Safety objective

  * To evaluate the safety and tolerability of Trastuzumab deruxtecan.(AEs/SAEs, Vital signs, Collection of clinical chemistry/haematology parameters, ECGs) 2. Exploratory Purpose
  * To identify mechanisms of adaptive resistance using Guardant 360 panel. To conduct NGS using Guardant 360 panel in serial plasma collection before treatment and at the time of progression.
  * To identify the profiling of interstitial lung disease (ILD) after treatment of T-DXd. To perform the baseline and follow-up PFT. To perform high-resolution chest CT to evaluate for ILD by radiologic expert. To evaluate cytokine level in serially collected plasma (every 6 weeks for the first 24 weeks and then every 12 weeks). The investigators recommend doing one HRCT at baseline and a second one in the event of ILD.

    3. Background Human epidermal growth factor receptor 2 (HER2, ERBB2)-activating mutations occur in 2% of lung cancers as a distinct molecular target. HER2-targeted therapy is standard of care for HER2-mutation positive non-small cell lung cancer (NSCLC).

Trastuzumab deruxtecan (T-DXd, DS-8201, Enhertu) is a novel antibody drug conjugate that is comprised of 3 components: a humanized anti-HER2 IgG1 monoclonal antibody with the same amino acid sequence as trastuzumab; a topoisomerase I inhibitor payload, an exatecan derivative; and a tetrapeptide-based cleavable linker.

Recently, T-DXd induced a confirmed objective response rate (ORR) of almost 61% and a durable benefit in heavily pre-treated patients with advanced HER2-positive breast cancer, according to results from the phase II DESTINY-Breast01 trial. In addition, the DESTINY-Gastric trial showed the superiority of T-DXd compared with standard chemotherapy in terms of response rate and progression-free and overall survival in this setting. Altogether, T-DXd received breakthrough therapy designation and orphan drug designation in gastric cancer, and approval for the treatment of advanced HER2-positive breast cancer. Recently, T-DXd showed durable systemic disease control along with CNS response. Ongoing trials are assessing the activity of T-DXd in patients with breast cancer and active brain metastases.

T-DXd has been approved in the US for the treatment of adult patients with unresectable or metastatic NSCLC whose tumours have activating HER2 mutations, as detected by a FDA-approved test, and who have received a prior systemic therapy. The accelerated approval by the FDA was based on the results from the DESTINY-Lung02 Phase II trial. An interim efficacy analysis in a pre-specified patient cohort showed T-DXd (5.4mg/kg) demonstrated a confirmed ORR of 57.7% (n=52; 95% CI 43.2-71.3), as assessed by blinded independent central review, in patients with previously treated unresectable or metastatic non-squamous HER2-mutant NSCLC. Complete responses (CR) were seen in 1.9% of patients and partial responses (PR) in 55.8% of patients with a median DoR of 8.7 months (95% CI 7.1-NE).

DETAILED DESCRIPTION:
4. Hypothesis T-DXd is actually approved for previously treated HER2m metastatic NSCLC patients but there is a gap of knowledge about intracranial response on T-DXd in NSCLC patients with brain metastasis. Therefore, in this study, the investigators aim to focus on the intracranial treatment outcome in HER2 mut NSCLC patients with brain metastasis.

Additionally, T-DXd has been shown to harbor more efficacy in HER2-mutated patients rather than HER2-overexpressing NSCLC patients.

However, severe life-threatening interstitial lung disease (ILD), including pneumonitis, can occur in patients treated with T-DXd. A recent findings demonstrated that ILD occurred in less than 16% of patients with HER2-positive metastatic breast cancer following treatment with T-DXd. Although the majority of these cases were grade 1 or 2, ILD remains an important risk, which highlights the need for close monitoring and early identification of ILD. Several cytokines, which activate JAK/STAT pathway, such as IL-4, IL-13, IL-6, IL-11 and IL-31, are implicated in the pathogenicity of ILD. However, there is no prospective study which evaluated the association of cytokines with the onset of drug-induced ILD.

Given the activity of T-DXd in HER2-mutant lung cancer, the investigators hypothesized that HER2-mutated tumors harbor susceptibility to HER2 ADCs and designed this phase 2 clinical trial of T-DXd in NSCLC HER2-mutant patients with brain metastases.

5. Study procedure This is Phase 2, Single arm, multi-centres', Open labelled study to assess efficacy and safety of T-DXd in HER2-mutant advanced lung cancer patients with asymptomatic brain metastases.

Advanced or metastatic non-squamous NSCLC with HER2 mutation regardless of HER2 expression with asymptomatic brain metastasis at baseline will be treated with T-DXd every 3weeks.

* HER2 activating mutation is based on local assessment of archival tissue or plasma ctDNA analysis. HER2 activating mutation are included exon 19 or 20.
* For resistance mechanism analysis, the investigators plan to conduct serial plasma collection from patients receiving T-DXd (before treatment and at the time of progression) to identify mechanisms of adaptive resistance using Guardant 360 panel.
* To identify the profiling of interstial lung disease (ILD) after treatment of T-DXd, the investigators plan to perform the baseline and follow-up PFT. The high-resolution CT will be evaluated for ILD by radiologic expert. The investigators serially collected plama for evaluation of cytokine (every 6 weeks for the first 24 weeks and then every 12 weeks). Pulmonologist, expert for ILD, will involve the ILD management when the patients show the ILD pattern and the symptoms suspicious for ILD.

<Detailed Description>

1. Objective:

   * Primary objective

     - Median Intracranial Progression-free survival(icPFS) as defined by RANO(Response Assessment in Neuro-Oncology) criteria
   * Secondary objective

     * Progression free survival(PFS) as defined by RECIST 1.1
     * Median Intracranial progression free survival(icPFS) as defined by RECIST 1.1
     * Intracranial objective response rate(icORR) as defined by RECIST 1.1
     * Overall response rate(ORR) as defined by RECIST 1.1
     * Duration of response(DoR) as defined by RECIST 1.1
     * Disease control rate (DCR) defined by RECIST 1.1
     * Overall survival (OS) ; The time from the date of inital IP administration to death due to any cause
     * Pattern of Progression ; Site of next progression
   * Safety objective

     - To evaluate the safety and tolerability of Trastuzumab deruxtecan.(AEs/SAEs, Vital signs, Collection of clinical chemistry/haematology parameters, ECGs)
   * Exploratory Purpose

     * To identify mechanisms of adaptive resistance using Guardant 360 panel. To conduct NGS using Guardant 360 panel in serial plasma collection before treatment and at the time of progression.
     * To identify the profiling of interstitial lung disease (ILD) after treatment of T-DXd. To perform the baseline and follow-up PFT. To perform high-resolution chest CT to evaluate for ILD by radiologic expert. To evaluate cytokine level in serially collected plasma (every 6 weeks for the first 24 weeks and then every 12 weeks). We recommend doing one HRCT at baseline and a second one in the event of ILD.
2. Background Human epidermal growth factor receptor 2 (HER2, ERBB2)-activating mutations occur in 2% of lung cancers as a distinct molecular target. HER2-targeted therapy is standard of care for HER2-mutation positive non-small cell lung cancer (NSCLC).

   Trastuzumab deruxtecan (T-DXd, DS-8201, Enhertu) is a novel antibody drug conjugate that is comprised of 3 components: a humanized anti-HER2 IgG1 monoclonal antibody with the same amino acid sequence as trastuzumab; a topoisomerase I inhibitor payload, an exatecan derivative; and a tetrapeptide-based cleavable linker.

   Recently, T-DXd induced a confirmed objective response rate (ORR) of almost 61% and a durable benefit in heavily pre-treated patients with advanced HER2-positive breast cancer, according to results from the phase II DESTINY-Breast01 trial. In addition, the DESTINY-Gastric trial showed the superiority of T-DXd compared with standard chemotherapy in terms of response rate and progression-free and overall survival in this setting. Altogether, T-DXd received breakthrough therapy designation and orphan drug designation in gastric cancer, and approval for the treatment of advanced HER2-positive breast cancer. Recently, T-DXd showed durable systemic disease control along with CNS response. Ongoing trials are assessing the activity of T-DXd in patients with breast cancer and active brain metastases.

   T-DXd has been approved in the US for the treatment of adult patients with unresectable or metastatic NSCLC whose tumours have activating HER2 mutations, as detected by a FDA-approved test, and who have received a prior systemic therapy. The accelerated approval by the FDA was based on the results from the DESTINY-Lung02 Phase II trial. An interim efficacy analysis in a pre-specified patient cohort showed T-DXd (5.4mg/kg) demonstrated a confirmed ORR of 57.7% (n=52; 95% CI 43.2-71.3), as assessed by blinded independent central review, in patients with previously treated unresectable or metastatic non-squamous HER2-mutant NSCLC. Complete responses (CR) were seen in 1.9% of patients and partial responses (PR) in 55.8% of patients with a median DoR of 8.7 months (95% CI 7.1-NE).
3. Hypothesis T-DXd is actually approved for previously treated HER2m metastatic NSCLC patients but there is a gap of knowledge about intracranial response on T-DXd in NSCLC patients with brain metastasis. Therefore, in this study, we aim to focus on the intracranial treatment outcome in HER2 mut NSCLC patients with brain metastasis.

   Additionally, T-DXd has been shown to harbor more efficacy in HER2-mutated patients rather than HER2-overexpressing NSCLC patients.

   However, severe life-threatening interstitial lung disease (ILD), including pneumonitis, can occur in patients treated with T-DXd. A recent findings demonstrated that ILD occurred in less than 16% of patients with HER2-positive metastatic breast cancer following treatment with T-DXd. Although the majority of these cases were grade 1 or 2, ILD remains an important risk, which highlights the need for close monitoring and early identification of ILD. Several cytokines, which activate JAK/STAT pathway, such as IL-4, IL-13, IL-6, IL-11 and IL-31, are implicated in the pathogenicity of ILD. However, there is no prospective study which evaluated the association of cytokines with the onset of drug-induced ILD.

   Given the activity of T-DXd in HER2-mutant lung cancer, we hypothesized that HER2-mutated tumors harbor susceptibility to HER2 ADCs and designed this phase 2 clinical trial of T-DXd in NSCLC HER2-mutant patients with brain metastases.
4. Study procedure This is Phase 2, Single arm, multi-centres', Open labelled study to assess efficacy and safety of T-DXd in HER2-mutant advanced lung cancer patients with asymptomatic brain metastases.

Advanced or metastatic non-squamous NSCLC with HER2 mutation regardless of HER2 expression with asymptomatic brain metastasis at baseline will be treated with T-DXd every 3weeks.

* HER2 activating mutation is based on local assessment of archival tissue or plasma ctDNA analysis. HER2 activating mutation are included exon 19 or 20.
* For resistance mechanism analysis, we plan to conduct serial plasma collection from patients receiving T-DXd (before treatment and at the time of progression) to identify mechanisms of adaptive resistance using Guardant 360 panel.
* To identify the profiling of interstial lung disease (ILD) after treatment of T-DXd, we plan to perform the baseline and follow-up PFT. The high-resolution CT will be evaluated for ILD by radiologic expert. We serially collected plama for evaluation of cytokine (every 6 weeks for the first 24 weeks and then every 12 weeks). Pulmonologist, expert for ILD, will involve the ILD management when the patients show the ILD pattern and the symptoms suspicious for ILD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 or more than 20 years-old
2. Histologically confirmed, "locally advanced and unresectable NSCLC not amenable to treatment with curative intent (surgery or chemoradiotherapy) or recurrent or de novo-metastatic non-squamous NSCLC (according to Version 8 of the IASLC Staging Manual in Thoracic Oncology) locally advanced or metastatic non-squamous NSCLC (Participants with mixed histology are eligible if adenocarcinoma is the predominant histology).
3. Activating HER2-mutation documented by NGS in tissue or plasma (include activating HER2 mutation in exon 19 or 20, i.e. , Exon 20: A775_G776insYVMA insertion/duplication; point mutations, L755S and G776C; transmembrane and the juxtamembrane domains G660D, R678Q, E693K and Q709Ldocumented mutation) regardless of HER2 expression.

   HER2 expression on tissue based on IHC (IHC 1+, 2+, or 3+)
4. Asymptomatic brain metastases at baseline without local therapy for brain metastasis or stable brain metastasis after local therapy (WBRTx, SRS, GKS etc), which is defined as patients who are not requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
5. Prior failure on any systemic chemotherapy platinum-based chemotherapy
6. Measurable disease according to RECIST version 1.1Response Assessment in Neuro-Oncology Criteria (RANO)
7. LVEF ≥ 50% within 28 days before randomization/enrollmentfirst dose .
8. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1.
9. Adequate organ and bone marrow function within 14 days before randomization/enrolment first dose as described in Table 1 below. All parameters must meet the inclusion criteria on the same day, and must be the most recent results available.

   Table 1 Parameters for Adequate Organ and Bone Marrow Function Adequate bone marrow function Platelet Count ≥ 100000/mm3. Haemoglobin ≥ 9.0 g/dL Absolute neutrophil count ≥ 1500/mm3 Adequate hepatic function Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN (< 5×ULN in participants with liver metastases) Total Bilirubin ≤ 1.5×ULN if no liver metastases or < 3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline Serum albumin ≥ 2.5 g/dL Adequate renal function CrCL ≥ 30 mL/min as determined by Cockcroft Gault (using actual body weight).

   Males:

   CLcr (mL/min) = "[140 - age (years)] × weight (kg)" /"72 × serum creatinine (mg/dL)"

   Females:

   (CLcr (mL/min) = "[140 - age (years)] × weight (kg)" /"72 × serum creatinine (mg/dL)" × 0.85 Adequate blood clotting function International normalised ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 × ULN

   *CrCL = calculated creatinine clearance; ULN = upper limit of normal
10. Adequate treatment washout period before enrollment, defined in Table 2 below:

    Table 2 Adequate treatment washout periods Treatment / Minimum Washout Period Major Surgery ≥ 4 weeks Radiation Therapy including palliative stereotactic radiation therapy to chest ≥ 4 weeks Palliative stereotactic radiation therapy to other anatomic areas including whole brain radiation, bone radiation and GKS ≥ 2 weeks Anti-Cancer chemotherapy [Immunotherapy (non-antibody based therapy)] ≥ 43 weeks Antibody based anti-cancer therapy ≥ 4 weeks Targeted agents and small molecules ≥ 242 weeks or 5 half-lives, whichever is longer TKIs approved for treatment of NSCLC ≥ 1 week.
    * baseline CT scan must be completed after discontinuation of TKI
11. Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test . prior to each administration of IMP.
12. Women of childbearing potential are defined as those who are not surgically sterile (i.e. underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal(Over 60 years old ). Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
13. Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception, presented in Table 3. from the time of screening and must agree to continue using such precautions for 7 months after the last dose of IMP. Not all methods of contraception are highly effective. Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable.
14. Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period, as described in Table 3. In addition, male patients should refrain from fathering a child, or freezing or donating sperm from the time of randomisation/enrolment, throughout the study and for 4 months after the last dose of IMP. Preservation of sperm should be considered prior to enrollment in this study.
15. Female subjects must not donate, or retrieve for their own use, ova from the time of randomization/enrolment and throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrollment in this study.

Exclusion Criteria:

1. Active brain metastases that require intervention
2. Leptomeningeal metastases
3. Systemic antitumor therapy within 28 days(Targeted therapy, ≥ 2 weeks or 5 half-lives) before initiation of T-DXd
4. Radiation therapy(excluding palliative stereotactic radiation therapy to chest) or gamma-knife surgery within 2weeks before initiation of T-DXd
5. Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
6. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Subjects with untreated but clinically inactive brain metastases may be included in the study. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment/randomization.
7. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 2 or baseline
8. Patients with a medical history of myocardial infarction (MI) within 6 months before enrolment, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV),
9. History of (non-infectious) ILD / pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
10. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.(Using for prophylactic antibiotics is allowed.)
11. Active primary immunodeficiency, known uncontrolled active HIV infection or active hepatitis B or C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1 Day 1. Subjects with past or resolved hepatitis B virus (HBV) infection who are anti-HBc positive (+) are eligible only if they are HBsAg negative (-).
12. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects should be tested for HIV prior to randomization/enrollment if required by local regulations or institutional review board (IRB)/ethics committee (EC).
13. Receipt of live, attenuated vaccine within 30 days prior to the first dose of trastuzumab deruxtecan. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of trastuzumab deruxtecan. Note: Participants, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of study intervention.
14. Clinically significant pleural effusion, ascites or pericardial effusion that requires drainage.(Stable
15. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.)
16. Any autoimmune, connective tissue or inflammatory disorders (e.g. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for patients who are included in the study.
17. Prior complete pneumonectomy
18. Known allergy or hypersensitivity to study treatment or any of the study drug excipients.
19. History of severe hypersensitivity reactions to other monoclonal antibodies.
20. Pregnant or breastfeeding female patients, or patients who are planning to become pregnant.
21. Multiple primary malignancies within 3 years, with the exception of

    * adequately resected non-melanoma skin cancer
    * curatively treated in-situ disease
    * other solid tumors curatively treated Procedures for withdrawal of incorrectly enrolled subjects see Section 3.4.
22. Prior use of targeted HER2 treatments, except for TKIs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Median Intracranial Progression-free survival(icPFS) as defined by RANO criteria | When all enrolled patients have completed 12 months of follow-up

SECONDARY OUTCOMES:
Progression free survival as defined by RECIST 1.1 | When all enrolled patients have completed 12 months of follow-up
Median Intracranial Progression-free survival as defined by RECIST 1.1 | When all enrolled patients have completed 12 months of follow-up
Intracranial objective response rate(icORR) as defined by RECIST 1.1 | When all enrolled patients have completed 12 months of follow-up
Overall response rate as defined by RECIST 1.1 | When all enrolled patients have completed 12 months of follow-up
Duration of response as defined by RECIST 1.1 | When all enrolled patients have completed 12 months of follow-up
Disease control rate as defined by RECIST 1.1 | When all enrolled patients have completed 12 months of follow-up
Overall survival (The time from the date of initial IP administration to death due to any cause) | When all enrolled patients have completed 12 months of follow-up
Site of progression of response as defined by RECIST 1.1 | When all enrolled patients have completed 12 months of follow-up
Number of paitents with AE based on CTCAE | When all enrolled patients have completed 12 months of follow-up
  To evaluate the safety and tolerability of Trastuzumab deruxtecan.(AEs/SAEs, Vital signs, Collection of clinical chemistry/haematology parameters, ECGs)

CONTACTS AND LOCATIONS:
Overall Officials: Hye Ryun Kim, Principal Investigator — Yonsei University Health system, Severance Hospital
Locations (1):
- Yonsei University Health system, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No